CLINICAL TRIAL: NCT02140073
Title: Research of Efficient Use of Omeprazole in Combination With Domperidone in Gastroesophageal Reflux Disease of Mild to Moderate Severity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Belarusian Medical Academy of Post-Graduate Education (Other)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OM2013
Record Dates: First submitted 2014-03-24; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-03

CONDITIONS: GERD
Keywords: GERD; Omez; Omez DSR; heartburn; esophagitis; omeprazole; omeprazole+domperidone
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Esophagitis | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- omeprazole+domperidone SR (Experimental): patients with GERD receive omeprazole 20mg + domperidone SR 30mg , 2 capsules in the morning
  Interventions: Drug: omeprazole
- omeprazole (Active Comparator): omeprazole 40mg in the morning
  Interventions: Drug: omeprazole+domperidone SR

INTERVENTIONS:
Drug: omeprazole+domperidone SR — omeprazole 20mg+domperidone SR 30mg, 2 capsules in the morning
  Other Names: Omez DSR
  Arms: omeprazole
Drug: omeprazole — 40mg in the morning
  Other Names: Omez
  Arms: omeprazole+domperidone SR

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and tolerability of omeprazole in combination with domperidone in GERD treatment for subsequent efficient pharmacotherapy of GERD.

Objectives of the trial To assess the efficacy of omeprazole in combination with domperidone regarding change of incidence and severity of clinical symptoms of GERD during 8 weeks of treatment To compare the efficacy of omeprazole in combination with domperidone regarding change of incidence and severity of clinical symptoms of GERD during 8 weeks of treatment To assess the efficacy of omeprazole in combination with domperidone regarding change of incidence and severity of endoscopic symptoms of GERD during 8 weeks of treatment To compare the efficacy of omeprazole in combination with domperidone regarding change of incidence and severity of endoscopic symptoms of GERD during 8 weeks of treatment To determine the efficiency and advantages of one GERD therapy considering efficacy, safety, and individual variance of patients' reactions

DETAILED DESCRIPTION:
Study design . Primary and secondary endpoints

Primary endpoint:

• reduced incidence and severity of heartburn after 8 weeks of treatment with Omez-DSR preparation in comparison with OMEZ preparation.

Secondary endpoints:

* reduced severity of heartburn estimated against visual analog scale after 8 weeks of treatment;
* incidence of events of heartburn after 4 and 8 weeks of treatment;
* proportion of patients with completely jugulated heartburn at the 4th and 8th weeks of treatment;
* number of days without heartburn after 4 weeks of treatment;
* proportion of patients with resolved esophagitis after 8 weeks of treatment in subjects with esophagitis at the time of enrollment.

Safety endpoints:

* incidence of adverse events in the group of patients who received at least one dose of the medicinal product after randomization;
* incidence of serious adverse events;
* incidence of severe adverse events;
* incidence of adverse events definitely caused by administration of the tested medicinal product.

Description of the trial planned By its design the trial will be a randomized open comparative parallel study.

Study flow chart:

Screening=>Randomization=>Group 1(Omez-DSR),Group 2(Omez) =>Treatment=>Monitoring

13.3. Phases of the trial:

1. Screening - preliminary selection of subjects according to clinical criteria; signing of informed consent; prescription and conduction of screening procedures; decision on inclusion/exclusion of subject from the trial on the grounds of the results of screening procedures according to inclusion/exclusion criteria.
2. Randomization - random distribution of subjects included into the trial into two groups: group 1 - treatment with tested Omez-DSR preparation, group 2 - treatment with the comparator Omez.
3. Treatment - patients receive either Omez-DSR preparation or Omez preparation in the prescribed regimen according to the randomization number. Treatment shall be ambulatory; patients shall visit research center through specified periods.
4. After the end of treatment patients shall return to their usual lifestyle, but they are monitored to assess the efficacy of the therapy conducted and to record adverse events.

Description of measures allowing reducing the bias factor Randomization Randomization at phase 2 shall be performed using the WinPepi statistical program, option Masking Partial masking shall be used. Assessment of endoscopic examination at week 8 of treatment shall be blinded; the specialist conducting endoscopy shall not know which therapy was used. Statistical analysis shall be performed after coding of subjects; and during analysis it shall not be known which of the groups is receiving Omez-DSR, and which one - Omez.

Description of treatment Medical preparations authorized in the Republic of Belarus shall be used in the trial: Omez-DSR and Omez.

Dosage Dosage shall be performed in accordance with label recommendations of Omez-DSR and Omez preparations. Dose of Omez shall be 2 capsules/day (40 mg of omeprazole). Dose of Omez-DSR shall be 2 capsules/day (40 mg of omeprazole and 60 mg of domperidone).

Regimen Medicinal preparations shall be prescribed after randomization. Group 1 or OM-DP: the subjects from this group shall be supplied the preparation enough for 8 weeks of treatment. Group 2 or OM: the subjects shall be supplied the preparation enough for 8 weeks.

Features of the phases of the trial

Signing of informed consent:Screening, Assessment of inclusion/exclusion criteria:Screening,Randomization Complaints Screening,Randomization,Week 8/End of treatment,Monitoring After 28 days

Past and present history: Screening,Randomization Drug history: Screening,Week 8/End of treatment, Monitoring After 28 days Physical examination: Screening,Randomization,Week 8/End of treatment, Monitoring After 28 days Height, weight measurement: Screening,Week 8/End of treatment, Monitoring After 28 days Survey against the GERD-Q scale (values of 7 scores): Screening,Week 8/End of treatment Distribution of diaries:Randomization Esophagogastroduodenoscopy: Screening,Week 8/End of treatment Pregnancy test: Screening Distribution of preparation:Randomization Recording of adverse events:Week 8/End of treatment, Monitoring After 28 days Compliance assessment:Week 8/End of treatment

ELIGIBILITY:
Criteria of inclusion of subjects

* desire to participate in the trial and ability to sign the informed consent;
* age above 18;
* gastroesophageal reflux disease, manifested in heartburn no less than twice a week prior to the 1st visit;
* use for the trial period of safe contraception methods for women of fertile age;
* results of ultrasonography (US) of abdominal cavity organs (ACO) performed in the last 6 months before the enrollment.

Criteria of non-inclusion refusal to undergo the endoscopic examination;

* gastroesophageal reflux disease with severe esophagitis (grade С or D against the Los Angeles classification);
* Barrett esophagus;
* pregnancy or lactation;
* administration of nonsteroidal antiinflammatory drugs (NSAIDs), aspirin, bisphosphonates, nitrates, calcium antagonists, proton pump inhibitors or Н2-blockers, prokinetics, clopidogrel;
* participation in other clinical trial;
* history of allergic reaction or intolerance of components of medicinal products;
* esophageal stricture;
* gastrectomy or gastric resection;
* malignant neoplasms in any location at present;
* alcohol abuse;
* severe cardiovascular or respiratory insufficiency;
* hepatic insufficiency;
* renal insufficiency.

Criteria of exclusion

* investigator's opinion on the necessity to exclude the patient for their own benefit;
* erroneous enrollment;
* investigator's decision to exclude the patient due to serious deviation from the trial program;
* serious adverse events (SAEs) including death (stating the date of death);
* adverse events (AEs) requiring monitoring and drug therapy;
* acute diseases or conditions which in the investigator's opinion require the patient to be excluded from the trial;
* administration during the trial of NSAIDs, aspirin, bisphosphonates, nitrates, calcium antagonists, proton pump inhibitors or Н2-blockers, prokinetics, antacids (except for the tested MP or the comparator MP) or the necessity for such treatment to be prescribed;
* positive pregnancy test (for women);
* patient's failure to appear for the visit;
* patient's refusal to continue the trial;
* intolerance of the tested MP or the comparator MP;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
change incidence of heartburn after 8 weeks of treatment with Omez-DSR preparation in comparison with OMEZ preparation | change from baseline incidence of heartburn after 8 weeks of treatment
  questionnaire
change severity of heartburn after 8 weeks of treatment with Omez-DSR preparation in comparison with OMEZ preparation | change from baseline severity of heartburn at 8 weeks
  questionnaire

SECONDARY OUTCOMES:
proportion of patients with completely jugulated heartburn | 4 and 8 weeks of treatment
  number of patients with completely jugulated heartburn after 4 weeks of treatment and 8 weeks of treatment
number of days without heartburn | 4 weeks of treatment
  questionnaire
proportion of patients with resolved esophagitis | after 8 weeks of treatment
  based on Esophagogastroduodenoscopy in subjects with esophagitis at the time of enrollment

OTHER OUTCOMES:
incidence of adverse events in the group of patients who received at least one dose of the medicinal product after randomization | 8 weeks of treatment
  questionnaire
incidence of serious adverse events | 8 weeks of treatment
  questionnaire
incidence of severe adverse events | 8 weeks of treatment
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yury Kh Marakhouski, Professor of Clinical Medicine, Principal Investigator — Belarusian Medical Academy of Post-Graduate Education
Locations (2):
- Belarus (2):
  - Gastroenterology and Nutrition Department. Byelorussian Medical Academy Postgraduate Education, Minsk
  - Mother and Child National Reaserch Centre, Minsk

REFERENCES:
- [Derived] Marakhouski KY, Karaseva GA, Ulasivich DN, Marakhouski YK. Omeprazole-Domperidone Fixed Dose Combination vs Omeprazole Monotherapy: A Phase 4, Open-Label, Comparative, Parallel Randomized Controlled Study in Mild to Moderate Gastroesophageal Reflux Disease. Clin Med Insights Gastroenterol. 2017 May 31;10:1179552217709456. doi: 10.1177/1179552217709456. eCollection 2017. PMID 28607547